CLINICAL TRIAL: NCT03367923
Title: Step Into Wellness: A Program of Health and Recovery for Endometrial Cancer Survivors
Brief Title: Health and Recovery Program in Increasing Physical Activity Level in Stage IA-IIIA Endometrial Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-43094; NCI-2017-02149 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GYNEND0002 (Other: OnCore)
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cancer Survivor; Endometrial Carcinoma; Stage I Uterine Corpus Cancer AJCC v7; Stage IA Uterine Corpus Cancer AJCC v7; Stage IB Uterine Corpus Cancer AJCC v7; Stage II Uterine Corpus Cancer AJCC v7; Stage IIIA Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Counseling; Equipment and Supplies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (exercise counseling, Fitbit, phone call) (Experimental): Participants undergo an exercise counseling session at baseline and wear Fitbit tracker daily for 9 months. Participants receive a short phone call at 2, 4, 6, and 8 weeks, and at 4 and 5 months to discuss the average number of daily steps over the past 2 weeks and to encourage a goal of a 10% increase over the next 2-4 week time period.
  Interventions: Other: Counseling; Other: Fitbit tracker; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Telephone-Based Intervention
- Arm II (exercise counseling, Fitbit, email/text) (Experimental): Participants undergo an exercise counseling session at baseline and wear Fitbit tracker daily for 9 months. Participants receive an electronic communication (email/text) of their choice at 2, 4, 6, and 8 weeks, and at 4 and 5 months stating the average number of daily steps over the past 2 weeks and encouraging a goal of a 10% increase over the next 2-4 week time period.
  Interventions: Other: Communication Intervention; Other: Counseling; Other: Fitbit tracker; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Receive email/text
  Arms: Arm II (exercise counseling, Fitbit, email/text)
Other: Counseling — Undergo exercise counseling
  Other Names: Counseling Intervention
Other: Fitbit tracker — Wear Fitbit tracker
  Other Names: Device
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive phone call
  Arms: Arm I (exercise counseling, Fitbit, phone call)

SUMMARY:
This randomized phase II trial studies how well a health and recovery program works in increasing physical activity level in stage IA-IIIA endometrial cancer survivors. Health and recovery program which includes exercise counseling, Fitbit tracker, and phone or email/text communication may increase the level of physical activity in endometrial cancer survivors and promote and maintain behavior change at a lower cost.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:I. Determine the increase in activity level per participant where the baseline average number of steps is recorded during week 0-2 will be compared to average step count recorded during week 20-28.SECONDARY OBJECTIVES:I. Determining the rate of patients who have achieved a 50% increase in activity level in each communication group (telephone versus [vs.] electronic).II. Demonstrate that the rate of patients who have achieved an increased activity level of 50% as compared to the patient's baseline in the electronic/email group is not inferior to the rate in the telephone group.III. Evaluate changes in body mass index (BMI), waist circumference, blood pressure and pulse for the whole group, by communication group (electronic vs. telephone), and by activity level.IV. Evaluate the changes in quality of life, as assessed by Functional Assessment of Cancer Therapy-General (FACT-G), during the course of the study for the whole group, between the two groups (electronic vs. telephone), and based on activity level.V. Evaluate maintenance of activity level at 9 month (m) (week 32-40) (comparison activity level 9 m vs. 6 m) for the whole group, by group (electronic vs. telephone), and by activity level.OUTLINE: Patients are randomized to 1 of 2 arms.ARM I: Participants undergo an exercise counseling session at baseline and wear Fitbit tracker daily for 9 months. Participants receive a short phone call at 2, 4, 6, and 8 weeks, and at 4 and 5 months to discuss the average number of daily steps over the past 2 weeks and to encourage a goal of a 10% increase over the next 2-4 week time period.ARM II: Participants undergo an exercise counseling session at baseline and wear Fitbit tracker daily for 9 months. Participants receive an electronic communication (email/text) of their choice at 2, 4, 6, and 8 weeks, and at 4 and 5 months stating the average number of daily steps over the past 2 weeks and encouraging a goal of a 10% increase over the next 2-4 week time period.

ELIGIBILITY:
Inclusion Criteria:

* Stage IA-IIIA endometrial cancer patients with pathology reviewed at Stanford
* Patients must have undergone surgery as a part of their treatment for their endometrial cancer
* At least 3 months post treatment
* BMI > 25
* Life expectancy of at least one year
* Able to perform physical activity of walking
* Possession of a computer and/or smart phone and/or smart tablet
* Must be English or Spanish speaking

Exclusion Criteria:

* Other active cancer
* Receiving chemotherapy or other active treatment
* BMI < 60
* Diagnosis of uterine serous carcinoma or uterine sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Increase in activity level measured using Fitbit tracker | Up to week 20-28
  The increase in activity level will be determined where the baseline average number of steps recorded per patient during week 0 - 2 will be compared to the average step count recorded during week 20 - 28. The baseline measurement will be defined as the average step count reported by the patient during 0-2 weeks. At each subsequent time point the average step count per patient will be the average of the step counts recorded during the 2-4 weeks prior to the follow up visit. The average step count measured at 20-28 weeks will be compared to the baseline in a paired t test. The paired t test will

SECONDARY OUTCOMES:
Body mass index (BMI) | Up to 9 months
  BMI will be measured using the participant weight in kilograms over height (in meters) squared. Changes in BMI over time will be evaluated in a repeated measures model allowing for within patient correlation. The relationship between average step count and the BMI will be evaluated in a repeated measures model allowing for within patient correlation. Determining if there is a difference between the two groups in the relationship between step count and health measures outcome: BMI will also be evaluated in a repeated measures model allowing for within patient correlation.
Pulse | Up to 9 months
  Pulse will be measured using an automated cuff while the participant is sitting. Changes in pulse over time will be evaluated in a repeated measures model allowing for within patient correlation.
Blood pressure | Up to 9 months
  Blood pressure will be measured using an automated cuff while the participant is sitting. Changes in blood pressure over time will be evaluated in a repeated measures model allowing for within patient correlation.
Quality of life assessment using Functional Assessment of Cancer Therapy-General (FACT-G) | Up to 9 months
  The relationship between average step count and quality of life will be evaluated in a repeated measures model allowing for within patient correlation. Determining if there is a difference between the two groups in the relationship between step count and quality of life will also be evaluated in a repeated measures model allowing for within patient correlation.
Rate of increased activity level measured using Fitbit tracker | Up to week 20-28
  For each patient, the average step count for the time period week 20 - 28 will be compared to the baseline (week 0-2) average step count. If the increase in step count is 50% or more the patient will have achieved an increased activity level. The proportion of patients who have achieved an increased activity level will be calculated for each arm.
Rate of increased activity level measured using Fitbit tracker | Up to 9 months
  For each patient, the average step count for the time period 6 months (weeks 20-28) will be compared to the baseline average step count. Likewise, for each patient the average step count for the time period 9 months (weeks 32-40) will be compared to the baseline average step count. The proportion of patients who have achieved an increased activity level will be calculated for each arm at each time period 6 months and 9 months.
Waist circumference | Up to 9 months
  Waist circumference will be measured in centimeters at the level of the belly button while participant is standing. Changes in waist circumference over time will be evaluated in a repeated measures model allowing for within patient correlation. The relationship between average step count and the outcomes of: waist circumference will be evaluated in a repeated measures model allowing for within patient correlation. Determining if there is a difference between the two groups in the relationship between step count and health measures outcomes: waist circumference will also be evaluated in a repea

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, School of Medicine, Palo Alto, California
  - Stanford Cancer Center South Bay, San Jose, California